CLINICAL TRIAL: NCT02780518
Title: Airvo/Optiflow High Flow Nasal Oxygenation During Microlaryngeal Surgery - Assessing Effectiveness of Oxygenation and Carbon Dioxide Clearance
Brief Title: Airvo/Optiflow High Flow Nasal Oxygenation During Microlaryngeal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Airvo 2 not suitable for CO2 clearance, awaiting Optiflow THRIVE machine
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1605 Airvo Optiflow
Record Dates: First submitted 2016-05-12; First posted 2016-05-23 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Throat Disorders
Keywords: oxygen; carbon dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Airvo (Experimental): All patients scheduled for elective microlaryngeal surgery under general anaesthesia and subglottic high frequency jet ventilation
  Interventions: Device: Airvo

INTERVENTIONS:
Device: Airvo — Applying high flow nasal oxygen

SUMMARY:
Optiflow high flow nasal cannula (HFNC) oxygenation is a technique to provide oxygen to patients when they are paralysed under general anaesthesia. Their lungs are not moving, but the high flow allows oxygen to travel into their lungs. This is called 'apnoeic ventilation'. The investigators will be using this for patients undergoing surgery for their throat.

DETAILED DESCRIPTION:
Hypothesis:

Optiflow high flow nasal cannula (HFNC) oxygenation is a suitable technique for oxygenation and ventilation (apnoeic ventilation) for patients undergoing microlaryngeal surgery.

Aims:

1. Measure continuous pulse oximetry (oxygenation) and intermittent subglottic catheter sampling of end tidal carbon dioxide levels (ventilation) in the distal trachea during HFNC oxygenation
2. Measure intra-tracheal airway pressure during HFNC oxygenation

Methodology:

As a pilot study, the investigators will recruit up to 20 patients within a 12 month period scheduled for elective microlaryngeal surgery and high frequency jet ventilation. Standard monitoring and standard conduct of anaesthesia will be carried out: induction of general anaesthesia, insertion of a narrow catheter into the trachea and insertion of laryngeal mask airway. In addition, the study device (HFNC) will be placed into the entrance of the patient's nostrils. After removal of the laryngeal mask, HFNC oxygenation will commence. A surgical suspension laryngoscope will be inserted for microlaryngeal surgery (standard technique). The investigators will measure the adequacy of gas exchange, during of HFNC oxygenation and complications (cardiovascular, airway and respiratory). Data will be stored on a secure REDCap (Research Electronic Data Capture) system.

Importance:

HFNC oxygenation is a novel technique that depends on apnoeic oxygenation. Even though the patient is paralysed and not breathing, oxygenation and carbon dioxide clearance still occurs. This is due to the difference between the alveolar rates of oxygen removal and carbon dioxide excretion which generates a negative pressure gradient. Oxygenation of the patient is therefore due to the high inspiratory fraction of oxygen, apnoeic ventilation and the small continuous positive airway pressure caused by the high flow of gas. This pressure increases lung volume and recruits collapsed alveoli. Carbon dioxide clearance is due to gas mixing and flushing of the airway dead space. The additional humidification of the high flow oxygen prevents mucociliary damage of the airway.

HFNC has been shown beneficial in pre-oxygenation, oxygenation after extubation, and in the treatment of respiratory failure and heart failure. New uses in difficult airway management are now emerging. However, the main case series of HFNC use in difficult airways did not measure intra-operative airway pressures end tidal oxygen and carbon dioxide; these gases were only measured at the end of surgery and when a definitive airway was inserted. As far as the investigators are aware, there are no data on intra-operative, intra-tracheal airway pressures or oxygen or carbon dioxide during HFNC oxygenation. Our study aim is to fill this knowledge gap.

Potential benefits and risks:

The use of HFNC removes obstacles form the surgical field and this may make surgery easier and quicker to perform. Risks include: failed gas exchange, but this is minimized by abandoning HFNC oxygenation and instituting tracheal catheter jet ventilation via the in situ jet catheter (standard practice).

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective microlaryngeal surgery requiring general anaesthesia and jet ventilation. They must have a physical status of the American Society of Anesthesiologists (ASA) grade I/II and age 21 years or older.

Exclusion Criteria:

1. Patients with history of previous difficult endotracheal intubation
2. Patients with two or more predictors of difficult mask ventilation or difficult intubation or the combination of both
3. Patients with ASA grading of III and above are excluded from the study
4. Patients needing a rapid sequence induction for rapid securement of the airway
5. Pregnant women
6. Patients below the age of 21 years old
7. Patients unfit to give consent
8. Patients with nasal or sinus disease or problems
9. Patients with infective laryngeal disease e.g. papillomatosis

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with inadequate oxygenation as measured by pulse oximetry (SpO2<94%). | 30 minutes
  Continuous pulse oximetry will be monitored for participants during the study.

SECONDARY OUTCOMES:
Number of patients with inadequate carbon dioxide clearance (end tidal CO2>55 mmHg) | 30 minutes
  End tidal carbon dioxide will be measured by the sublgottic catheter already in situ in the trachea by continuous passive sampling and by intermittent low frequency jet ventilation
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 30 minutes
  The investigator will report the number of participants wtih adverse events that are related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wong, MBBS FRCA, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645